CLINICAL TRIAL: NCT07033767
Title: Exploring a Natural Solution for Childhood Obesity
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Western University (Other)
Collaborators: Western University, Canada (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Marina Ybarra, MD, MSc - Assistant Professor, Western University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 125367
Record Dates: First submitted 2025-06-10; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Children
Keywords: genistein; childhood obesity; children
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm study (Other): Arm Type: Single Group Assignment
  Assigned Intervention:
  Drug: Genistein
  Participants will receive genistein at 10-15 mg/kg/day (max 1500 mg/day) for the first 3 months.
  From months 3 to 6, the dose will be increased to 20-25 mg/kg/day (max 1500 mg/day).
  Genistein will be provided as 250 mg capsules. Capsules may be swallowed whole or opened and mixed with food or a beverage for those unable to swallow pills.
  Interim evaluations will be conducted at 3 and 6 months to assess tolerability, adherence, and efficacy.
  A post-treatment follow-up at 9 months (after a 3-month washout) will assess delayed adverse effects and the persistence of benefits after genistein discontinuation.
  Other Names:
  Sophora japonica extract
  Genistin (active metabolite)
  Interventions: Drug: genistein

INTERVENTIONS:
Drug: genistein — Participants will receive genistein treatment (10-15 mg/kg/day with a maximum dose of 1500mg/day) for 3 months. From the 3-month- to 6-month follow-up, participants will receive a dose of 20-25 mg/kg/day (with a maximum dose of 1500mg/day). According to participant preference, Genistein will be provided as a capsule (250mg per capsule). For participants that are unable to swallow the capsule the capsule may be opened and the powder from the capsule can be mixed with a beverage or food. Interim clinical evaluations will occur at 3 and 6 months to assess, tolerability, adherence and efficacy.. Post-treatment assessment after a 3-month washout will occur at 9 months to determine delayed adverse effects and persistence of beneficial effects after genistein discontinuation.

SUMMARY:
This study aims to assess the safety tolerability, adherence and effectiveness of genistein as an anti-obesity treatment for children and adolescents. The primary goal is determining how well genistein is tolerated and adhered to by pediatric patients with obesity. Secondary goals include evaluating its impact on body mass index z-scores and cardiometabolic risk factors, such as inflammation.

Participants aged 4-18 will be recruited from the Paediatric HEAL (Healthy Eating, Activity & Lifestyle) Program at the Children's Hospital - London Health Science Center in London, Ontario. They will receive genistein treatment over 6 months, with interim assessments at 3 and 6 months to monitor efficacy, safetytolerability, and adherence, and efficacy, and potentially increase the dose at the 3-month visit. A final assessment will occur after a 3-month washout to observe any lasting effects.

Blood and urine samples will be collected to analyze various adherence and health markers, including inflammatory and cardiometabolic factors. For participants who are of childbearing potential and have had their first menses, the blood analysis will also include pregnancy testing. Laboratory testing will be performed at baseline, at three and six months while taking genistein and three months after the washout period. Urine samples will also confirm that genistein has been taken appropriately throughout the study.

The study expects that genistein will be well-tolerated by children, reduce BMI z-scores by 0.2 (0.5), and improve cardiometabolic risk factors such as blood pressure, lipid profiles, and inflammation. A sample size of 60 participants has been calculated to achieve statistically significant results, which will inform more extensive studies on genistein's potential for managing pediatric obesity.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 4-17 years.
* Obesity defined as a BMI z-score ≥ 2 for age and sex, based on World Health Organization (WHO) reference standards.
* Stable or increasing BMI after at least 3 months of enrollment in the HEAL program.
* Inclusion of participants from all backgrounds, consistent with principles of equity, diversity, and inclusion.
* Participants and families who do not speak or read English will be included, provided interpreter services are available at LHSC's Children's Hospital.
* Participants who decline to enroll will continue receiving standard care in the HEAL program.

Exclusion Criteria:

* Known allergy to Sophora japonica (source of genistein).
* Diagnosis of type 2 diabetes (these patients are followed in a separate Diabetes Clinic).
* Current use of medications that may confound study outcomes, including:
* GLP-1 receptor agonists (e.g., Saxenda, Wegovy)
* ADHD medications (e.g., Concerta, Vyvanse, Abilify)
* Antipsychotic medications (e.g., Risperidone)
* Currently pregnant, breastfeeding, or planning to become pregnant during the study period.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) z-score | 6 months
  To assess the impact of genistein on Body Mass Index (BMI) z-scores, calculated using the World Health Organization (WHO) growth reference standards for age and sex.
  Scale: WHO BMI-for-age z-score
  Score Range: Typically from approximately -3 to +5
  Interpretation: Higher scores indicate greater degrees of obesity, and lower scores indicate improvement in weight status relative to age and sex norms.

SECONDARY OUTCOMES:
Tolerability of Genistein Treatment | 6 months
  To assess the tolerability of genistein as an anti-obesity treatment in children aged 4-18 years with obesity, as measured by the incidence of adverse events, treatment discontinuation rates, and tolerability questionnaires completed by caregivers and participants (e.g., Likert scale or standardized adverse event checklist).
Adherence to Genistein Treatment | 6 months
  To assess adherence to genistein as an anti-obesity treatment in children aged 4-18 years with obesity, as measured by the percentage of prescribed doses taken, recorded through pill counts, caregiver-reported adherence logs, and/or electronic medication monitoring (e.g., MEMS caps).

OTHER OUTCOMES:
Change in Fasting Glucose Levels | 6 months
  To assess the effect of genistein on fasting glucose levels, measured in mmol/L via standard clinical laboratory testing.
Change in Fasting Insulin Levels | 6 months
  To assess the effect of genistein on fasting insulin levels, measured in pmol/L via standard clinical laboratory testing.
Change in HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) | 6 months
  To assess insulin resistance using HOMA-IR, calculated from fasting insulin and glucose levels. Higher scores indicate greater insulin resistance.
  Unit of Measure: HOMA-IR index (unitless)
Change in Lipid Profile - Total Cholesterol | 6 months
  To assess changes in total cholesterol levels, measured in mmol/L via clinical laboratory tests.
Change in Lipid Profile - LDL-C | 6 months
  To assess changes in low-density lipoprotein cholesterol (LDL-C), measured in mmol/L.
Change in Lipid Profile - HDL-C | 6 months
  To assess changes in high-density lipoprotein cholesterol (HDL-C), measured in mmol/L.
Change in Lipid Profile - Triglycerides | 6 months
  To assess changes in triglyceride levels, measured in mmol/L.
Change in High-Sensitivity C-Reactive Protein (hs-CRP) | 6 months
  To assess inflammation using hs-CRP levels, measured in mg/L via standard blood test.
Change in Systolic and Diastolic Blood Pressure | 6 months
  To assess blood pressure changes using manual or automated blood pressure cuffs appropriate for pediatric populations. Reported in mmHg for both systolic and diastolic readings.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Ybarra, MD, MSc, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No
This is a single center study with only one primary investigator